CLINICAL TRIAL: NCT02729532
Title: Z 31411 - The Effect of Xpert MTB/RIF on Patient Health Outcomes and Empirical TB Treatment Among Persons Living With HIV/AIDS: A Parallel-Group Prospective Cohort Study Under Real-World Conditions in Lusaka, Zambia
Brief Title: Effect of Xpert MTB/RIF on Patient Outcomes
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-1697; US NIH Grant P30 AI50410-17 (Other Grant/Funding Number: US NIH)
Record Dates: First submitted 2016-01-05; First posted 2016-04-06 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Tuberculosis
Keywords: Extra-pulmonary tuberculosis; multiple drug resistant tuberculosis; mycobacterium tuberculosis; human immunodeficiency virus
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Extrapulmonary; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Xpert cohort: HIV-positive presumptive TB patients tested for TB using Xpert MTB/RIF assay (fluorescence microscopy and TB culture also done to serve as reference standard)
  Interventions: Device: Xpert
- Standard of Care cohort: HIV-positive presumptive TB patients tested for TB using standard of care testing (sputum smear microscopy plus clinical evaluation)

INTERVENTIONS:
Device: Xpert — The Xpert MTB/RIF assay is a nucleic acid amplification (NAA) test that uses a disposable cartridge with the GeneXpert Instrument System
  Other Names: Xpert MTB/RIF assay
  Groups: Xpert cohort

SUMMARY:
A parallel-group prospective cohort study among adult persons living with HIV/AIDS to study the effect of a new TB diagnostic test, Xpert MTB/RIF on: 1) TB case detection; 2) time to TB diagnosis and TB treatment; 3) presumptive TB patient drop-out from the TB diagnostic "cascade" before starting TB treatment; and 4) loss to follow-up after initiation of TB treatment.

DETAILED DESCRIPTION:
The Centre for Infectious Disease Research in Zambia (CIDRZ) in collaboration with the Zambian National TB Program (NTP) and the Ministry of Health (MOH) will provide near point-of-care Xpert testing at a high-volume anti-retroviral treatment (ART) clinic in Lusaka, Zambia. A total 892 study participants will be enrolled into two parallel cohorts-an "Xpert" and a "standard of care" (SOC) cohort over a 7-month period. The Xpert cohort will enrol participants at the health centre implementing Xpert. The SOC cohort will enrol participants from one health centre offering the standard of care (sputum smear microscopy plus clinical evaluation). A parallel-group prospective cohort study will be conducted by following participants in one cohort from each site for 210 days from the time of sputum submission, allowing sufficient person-time to observe all outcomes of interest, including completion of a standard course of ATT as well as patient drop-out and loss to follow-up.

A systematic facility assessment survey using an adapted version of the WHO Service Availability and Readiness Assessment tool will be conducted. Key informants will be interviewed.

ELIGIBILITY:
Inclusion Criteria:

* Able to spontaneously expectorate at least 2 sputum samples, in accordance with NTP guidelines
* Intend to continue receiving care at the respective study sites for at least 7 months
* Willing to provide locator information and allow contact by phone or home visit in the case of loss to follow up after initiating ATT

Exclusion Criteria:

* Received TB treatment within 60 days prior to enrolment and/or were diagnosed with TB within the last 6 months
* Cannot spontaneously expectorate sputum
* Are already enrolled in another study with might interfere with implementation of this study protocol
* Provided a sputum sample that results in a contaminated TB culture result

A key informant will be eligible for inclusion in the SARA facility survey component of the study if they meet the following criteria:

* 18 years of age or older
* clinic staff member at either Chilenje Health Centre or Chelstone Health Centre
* have previously been attached to, or are otherwise familiar with, departments offering HIV, TB and/or laboratory health services

Exclusion criteria:

-unwilling or unable to provide verbal informed consent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult presumptive TB patients 18 years or older with documented HIV-positive sero-status presenting for routine HIV care at two health centres in Lusaka, Zambia.
Sampling Method: Probability Sample
Enrollment: 776 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Culture-positive patient drop-out before accessing treatment | From study enrolment through confirmed drop out date at or before 210-days post enrollment
  For both cohorts, the proportion of patients not started on TB treatment by 210 days post-enrolment will be assessed.

SECONDARY OUTCOMES:
Time to TB treatment | time in days from study enrolment to initiation of anti-TB therapy (ATT) (through 210 days post-enrolment)
Percentage of participants who receive TB treatment within 14 days of enrolment (effect of Xpert on the accuracy of TB diagnosis) | study enrolment to 14 days of enrolment
  sensitivity of empirical TB diagnosis and treatment will be defined as the percentage of participants who received TB treatment within 14 days of enrolment among all those with a positive culture but negative or unavailable result for SM (for the SOC cohort), or negative or unavailable SM plus Xpert (for the Xpert cohort)
Percentage of participants who did not receive TB treatment 14 days post-enrolment (effect of Xpert on the accuracy of TB diagnosis) | study enrolment to 14 days of enrolment
  the specificity of empirical treatment will be defined as the percentage of participants who did not receive TB treatment 14 days post-enrolment among all those with a negative culture and negative or unavailable result for SM (in the SOC cohort), or negative or unavailable result for SM plus Xpert (in the Xpert cohort)
Time to TB Diagnosis | average of 28 days
  The World Health Organization definition of a TB case will be used
Number of TB patients lost to follow-up | The number of patients will be measured as time in days from study enrolment to confirmed drop out (confirmed as failure noted at 3 and 6 month chart review)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Herce, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Chelstone and Chilenje Health Centres, Lusaka, Zambia

REFERENCES:
- [Background] Botha E, Den Boon S, Verver S, Dunbar R, Lawrence KA, Bosman M, Enarson DA, Toms I, Beyers N. Initial default from tuberculosis treatment: how often does it happen and what are the reasons? Int J Tuberc Lung Dis. 2008 Jul;12(7):820-3. PMID 18544210
- [Background] World Health Organization. (2013). Global tuberculosis report 2013. Geneva: WHO.
- [Background] Millen SJ, Uys PW, Hargrove J, van Helden PD, Williams BG. The effect of diagnostic delays on the drop-out rate and the total delay to diagnosis of tuberculosis. PLoS One. 2008 Apr 9;3(4):e1933. doi: 10.1371/journal.pone.0001933. PMID 18398459
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Background] Boehme CC, Nicol MP, Nabeta P, Michael JS, Gotuzzo E, Tahirli R, Gler MT, Blakemore R, Worodria W, Gray C, Huang L, Caceres T, Mehdiyev R, Raymond L, Whitelaw A, Sagadevan K, Alexander H, Albert H, Cobelens F, Cox H, Alland D, Perkins MD. Feasibility, diagnostic accuracy, and effectiveness of decentralised use of the Xpert MTB/RIF test for diagnosis of tuberculosis and multidrug resistance: a multicentre implementation study. Lancet. 2011 Apr 30;377(9776):1495-505. doi: 10.1016/S0140-6736(11)60438-8. Epub 2011 Apr 18. PMID 21507477
- [Background] Lawn SD, Brooks SV, Kranzer K, Nicol MP, Whitelaw A, Vogt M, Bekker LG, Wood R. Screening for HIV-associated tuberculosis and rifampicin resistance before antiretroviral therapy using the Xpert MTB/RIF assay: a prospective study. PLoS Med. 2011 Jul;8(7):e1001067. doi: 10.1371/journal.pmed.1001067. Epub 2011 Jul 26. PMID 21818180
- [Background] Boehme, C. C. Oral Presentation, 20th Conference on Retroviruses and Opportunistic Infections. Georgia World Conference Centre, Atlanta, USA, March 3-6, 2013.
- [Background] Theron G, Zijenah L, Chanda D, Clowes P, Rachow A, Lesosky M, Bara W, Mungofa S, Pai M, Hoelscher M, Dowdy D, Pym A, Mwaba P, Mason P, Peter J, Dheda K; TB-NEAT team. Feasibility, accuracy, and clinical effect of point-of-care Xpert MTB/RIF testing for tuberculosis in primary-care settings in Africa: a multicentre, randomised, controlled trial. Lancet. 2014 Feb 1;383(9915):424-35. doi: 10.1016/S0140-6736(13)62073-5. Epub 2013 Oct 28. PMID 24176144
- [Background] Office of the U.S. Global AIDS Coordinator. Scaling Up TB Prevention, Screening, Diagnosis and Care in Zambia: Implementing the WHO 3I's, Program Protocol. Lusaka: Centers for Disease Control and Prevention-Zambia, 2012.
- [Background] Kivihya-Ndugga LE, van Cleeff MR, Githui WA, Nganga LW, Kibuga DK, Odhiambo JA, Klatser PR. A comprehensive comparison of Ziehl-Neelsen and fluorescence microscopy for the diagnosis of tuberculosis in a resource-poor urban setting. Int J Tuberc Lung Dis. 2003 Dec;7(12):1163-71. PMID 14677891
- [Background] UNAIDS. Global Report: UNAIDS report on the global AIDS epidemic 2013. Geneva: Joint United Nations Programme on HIV/AIDS, 2013.
- [Background] Getahun H, Harrington M, O'Brien R, Nunn P. Diagnosis of smear-negative pulmonary tuberculosis in people with HIV infection or AIDS in resource-constrained settings: informing urgent policy changes. Lancet. 2007 Jun 16;369(9578):2042-2049. doi: 10.1016/S0140-6736(07)60284-0. PMID 17574096
- [Background] Steingart KR, Henry M, Ng V, Hopewell PC, Ramsay A, Cunningham J, Urbanczik R, Perkins M, Aziz MA, Pai M. Fluorescence versus conventional sputum smear microscopy for tuberculosis: a systematic review. Lancet Infect Dis. 2006 Sep;6(9):570-81. doi: 10.1016/S1473-3099(06)70578-3. PMID 16931408
- [Background] Sreeramareddy CT, Panduru KV, Menten J, Van den Ende J. Time delays in diagnosis of pulmonary tuberculosis: a systematic review of literature. BMC Infect Dis. 2009 Jun 11;9:91. doi: 10.1186/1471-2334-9-91. PMID 19519917
- [Background] Cohen T, Murray M, Wallengren K, Alvarez GG, Samuel EY, Wilson D. The prevalence and drug sensitivity of tuberculosis among patients dying in hospital in KwaZulu-Natal, South Africa: a postmortem study. PLoS Med. 2010 Jun 22;7(6):e1000296. doi: 10.1371/journal.pmed.1000296. PMID 20582324
- [Background] Vassall A, van Kampen S, Sohn H, Michael JS, John KR, den Boon S, Davis JL, Whitelaw A, Nicol MP, Gler MT, Khaliqov A, Zamudio C, Perkins MD, Boehme CC, Cobelens F. Rapid diagnosis of tuberculosis with the Xpert MTB/RIF assay in high burden countries: a cost-effectiveness analysis. PLoS Med. 2011 Nov;8(11):e1001120. doi: 10.1371/journal.pmed.1001120. Epub 2011 Nov 8. PMID 22087078
- [Background] Steingart KR, Sohn H, Schiller I, Kloda LA, Boehme CC, Pai M, Dendukuri N. Xpert(R) MTB/RIF assay for pulmonary tuberculosis and rifampicin resistance in adults. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD009593. doi: 10.1002/14651858.CD009593.pub2. PMID 23440842
- [Background] Dowdy DW, Davis JL, den Boon S, Walter ND, Katamba A, Cattamanchi A. Population-level impact of same-day microscopy and Xpert MTB/RIF for tuberculosis diagnosis in Africa. PLoS One. 2013 Aug 12;8(8):e70485. doi: 10.1371/journal.pone.0070485. eCollection 2013. PMID 23950942
- [Background] Van Rie A, Page-Shipp L, Hanrahan CF, Schnippel K, Dansey H, Bassett J, Clouse K, Scott L, Stevens W, Sanne I. Point-of-care Xpert(R) MTB/RIF for smear-negative tuberculosis suspects at a primary care clinic in South Africa. Int J Tuberc Lung Dis. 2013 Mar;17(3):368-72. doi: 10.5588/ijtld.12.0392. PMID 23407225
- [Background] Hanrahan CF, Selibas K, Deery CB, Dansey H, Clouse K, Bassett J, Scott L, Stevens W, Sanne I, Van Rie A. Time to treatment and patient outcomes among TB suspects screened by a single point-of-care xpert MTB/RIF at a primary care clinic in Johannesburg, South Africa. PLoS One. 2013 Jun 6;8(6):e65421. doi: 10.1371/journal.pone.0065421. Print 2013. PMID 23762367
- [Background] Clouse K, Page-Shipp L, Dansey H, Moatlhodi B, Scott L, Bassett J, Stevens W, Sanne I, Van Rie A. Implementation of Xpert MTB/RIF for routine point-of-care diagnosis of tuberculosis at the primary care level. S Afr Med J. 2012 Sep 7;102(10):805-7. doi: 10.7196/samj.5851. PMID 23034211
- [Background] Lawn SD, Ayles H, Egwaga S, Williams B, Mukadi YD, Santos Filho ED, Godfrey-Faussett P, Granich RM, Harries AD. Potential utility of empirical tuberculosis treatment for HIV-infected patients with advanced immunodeficiency in high TB-HIV burden settings. Int J Tuberc Lung Dis. 2011 Mar;15(3):287-95. PMID 21333094
- [Background] Yoon C, Cattamanchi A, Davis JL, Worodria W, den Boon S, Kalema N, Katagira W, Kaswabuli S, Miller C, Andama A, Albert H, Nabeta P, Gray C, Ayakaka I, Huang L. Impact of Xpert MTB/RIF testing on tuberculosis management and outcomes in hospitalized patients in Uganda. PLoS One. 2012;7(11):e48599. doi: 10.1371/journal.pone.0048599. Epub 2012 Nov 6. PMID 23139799
- [Background] Global Health Workforce Statistics, World Health Organization, Geneva. Accessed online at: http://www.who.int/hrh/statistics/hwfstats/ on November 24, 2013.
- [Background] WHO. Guidelines for intensified tuberculosis case-finding and isoniazid preventative therapy for people living with HIV in resource-constrained settings. Geneva: World Health Organization, 2011.
- [Background] Treatment of Tuberculosis: Guidelines. 4th edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138748/ PMID 23741786
- [Background] Global Laboratory Initiative. Laboratory diagnosis of tuberculosis by sputum microscopy: The handbook. Geneva: Global Laboratory Initiative, 2013.
- [Background] Joffe MM, Rosenbaum PR. Invited commentary: propensity scores. Am J Epidemiol. 1999 Aug 15;150(4):327-33. doi: 10.1093/oxfordjournals.aje.a010011. PMID 10453808
- [Background] WHO/TDR/FIND. Diagnostics for tuberculosis: Global demand and market potential. Geneva: World Health Organization, 2006.
- [Background] Balcha TT, Sturegard E, Winqvist N, Skogmar S, Reepalu A, Jemal ZH, Tibesso G, Schon T, Bjorkman P. Intensified tuberculosis case-finding in HIV-positive adults managed at Ethiopian health centers: diagnostic yield of Xpert MTB/RIF compared with smear microscopy and liquid culture. PLoS One. 2014 Jan 22;9(1):e85478. doi: 10.1371/journal.pone.0085478. eCollection 2014. PMID 24465572
- [Background] Theron G, Peter J, Dowdy D, Langley I, Squire SB, Dheda K. Do high rates of empirical treatment undermine the potential effect of new diagnostic tests for tuberculosis in high-burden settings? Lancet Infect Dis. 2014 Jun;14(6):527-32. doi: 10.1016/S1473-3099(13)70360-8. Epub 2014 Jan 15. PMID 24438820
- [Background] Conwell DS, Mosher A, Khan A, Tapy J, Sandman L, Vernon A, Horsburgh CR Jr. Factors associated with loss to follow-up in a large tuberculosis treatment trial (TBTC Study 22). Contemp Clin Trials. 2007 May;28(3):288-94. doi: 10.1016/j.cct.2006.09.003. Epub 2006 Sep 28. PMID 17107825
- [Background] Henostroza G, Harris J, Siyambango M, et al. High prevalence of tuberculosis among new HIV care enrolees in Zambia: urgent need for an enhanced screening approach. Oral presentation, 43rd World Conference on Lung Health. Kuala Lumpur Convention Centre, Kuala Lumpur, Malaysia. November 13 - 17, 2012.
- [Background] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648
- [Background] Chang K, Lu W, Wang J, Zhang K, Jia S, Li F, Deng S, Chen M. Rapid and effective diagnosis of tuberculosis and rifampicin resistance with Xpert MTB/RIF assay: a meta-analysis. J Infect. 2012 Jun;64(6):580-8. doi: 10.1016/j.jinf.2012.02.012. Epub 2012 Feb 27. PMID 22381459
- [Background] Moure R, Martin R, Alcaide F. Effectiveness of an integrated real-time PCR method for detection of the Mycobacterium tuberculosis complex in smear-negative extrapulmonary samples in an area of low tuberculosis prevalence. J Clin Microbiol. 2012 Feb;50(2):513-5. doi: 10.1128/JCM.06467-11. Epub 2011 Dec 7. PMID 22162564
- [Background] Ministry of Health, Republic of Zambia. Managing Tuberculosis in the HIV Setting in Zambia. Lusaka: Ministry of Health, 2014.
- See also: University of North Carolina website — http://www.unc.edu